CLINICAL TRIAL: NCT04467216
Title: Virtual Reality Motor-cognitive Training for Older People With Cognitive Frailty: A Pilot Trial
Brief Title: VR Motor-cognitive Training for Cognitive Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Rick Kwan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZB1H
Record Dates: First submitted 2020-06-11; First posted 2020-07-10 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Frailty
Keywords: Cognitive frailty; Motor-cognitive training; Virtual reality; Gamification

STUDY DESIGN:
Intervention Model Description: A total of 16 subjects with cognitive frailty will be assigned into 2 groups. Eight participants will be assigned to the intervention group in which they will undertake VR simultaneous motor-cognitive training and eight participants will be assigned to the control group in which existing forms of non-VR sequential motor-cognitive training will be provided.
  Both intervention and control groups will employ the same intervention dosage including course, session duration and frequency. The following dosage is employed because they are also the same dosage used in the VR simultaneous motor-cognitive training that we proposed. I.e.,
  * Course: eight weeks
  * Session duration: 30 minutes
  * Frequency: twice per week
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors at both pre- and post-observations will be blinded to the group label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This arm will undertake VR simultaneous motor-cognitive training in 30 minutes session, twice a week for 8 weeks
  Interventions: Device: Computerised cognitive training using virtual reality
- Control Group (No Intervention): This arm will be doing existing forms of motor-cognitive training in 30 minutes session, twice a week for 8 weeks

INTERVENTIONS:
Device: Computerised cognitive training using virtual reality — Immersive VR training system tailor-made for the daily living experiences in the Hong Kong context to provide interactive experiences for older people in Hong Kong.The VR systems available in the market for older people are only for non-interactive activities (e.g., watching movies) to provide unusual experiences for disabled older people who cannot travel too far from home.
  Arms: Intervention group

SUMMARY:
Cognitive frailty is a clinical syndrome in which cognitive impairment (e.g., poor memory, visuospatial function) and physical frailty (e.g., slowness, poor muscle strength, physical inactivity) co-exist. It is prevalent in community-dwelling older people. The progressive decline of cognitive and physical functions restricts older people from participating in activities (e.g., social get-togethers). Reduced participation further jeopardizes their life-space mobility (e.g., ability to travel to areas far away from home). Therefore, those with cognitive frailty are at risk of developing dementia and becoming dependent.

Simultaneous motor-cognitive training is more effective at promoting optimal functioning in older people than motor or cognitive training alone. Gaming is effective at promoting the motivation to participate. The contents of games in the market are unrelated to the context or daily living of the elderly. Currently, available training is non-simultaneous. This makes the training less transferable to the daily life of the elderly and reduces its effects.

Virtual reality (VR) technology can provide a virtual space that mimics the real environment. This allows clients to participate in daily activities in a virtual space. Older people can be trained to improve their cognitive and physical skills in a painless, fun way. However, the effect and feasibility of employing simultaneous motor-cognitive training launching on a VR platform mimicking the daily living environment in older people with cognitive frailty is poorly known. This pilot trial aims to examine the preliminary effects on cognitive function and frailty syndrome, as well as examine the feasibility.

DETAILED DESCRIPTION:
In the intervention, VR will be employed to simulate a daily living environment familiar to older people. Participants will wear a commercially available head-mounted VR system with hand-held controllers to experience the participation of daily activities in a virtual environment. Simultaneous physical and cognitive training will be embedded in the training system to promote optimal function. Participants will attend physical training in a sitting position through cycling on an ergometer and moving the hand-held controllers. Motion sensors built into the VR system and ergometer will track these movements to control everyday tasks in the virtual environment (e.g., moving around the city). Simultaneously, participants will undergo cognitive training by participating in various tasks demanding cognitive functions, such as visual-spatial (e.g., wayfinding) and problem-solving (e.g., wallet loss) functions. Gamification will be employed to promote the motivation to participate. All training activities will be gamified by blending in fun elements, such as difficulty-levelling, competition, and e-tokens. Co-participation is allowed to promote interpersonal interactions. The prototype enables real-time co-viewing among participants. Other elderly centre members and the activity facilitators can share the view of the participants in the game on either a large-screen monitor or a tablet computer. They can simultaneously talk about and share their gaming experiences.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 60 years,
2. Community dwelling, as defined by living at home without staying in long-term care facilities (e.g., nursing home) in the last 12 months, and
3. Cognitive frailty, as defined by co-existence of mild cognitive impairment and physical frailty,

   1. Mild cognitive impairment, measured by Montreal Cognitive Assessment (MoCA) ≤ 25 and Clinical Dementia Rating (CDR) = 0.5, and
   2. Frailty status from pre-frail to frail, measured by Fried Frailty Phenotype score ≥ 1.

Exclusion criteria

1. Diagnosed dementia, according to subjects' medical record, or
2. Probable dementia, as defined by MoCA ≤ 18, or
3. Mobility restriction, as defined by Modified Functional Ambulatory Classification (MFAC) < Category 7 (i.e., Outdoor walker), or

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Global cognitive function | Change is being assessed: "baseline" and "immediately after the completion" (2 months)
  Montreal Cognitive Assessment (score), scores on the MoCA range from zero to 30.
  With a score of 26 and higher generally considered normal, with 25 to 18 are considered Mild Cognitive Impairment and with score lower then 18 are defined as Alzheimer's disease.
Selective attention | Change is being assessed: "baseline" and "immediately after the completion" (2 months)
  Stroop test (score)
Visual-spatial perception | Change is being assessed: "baseline" and "immediately after the completion" (2 months)
  Visual Object Space Perception test (score)

SECONDARY OUTCOMES:
Frailty | Change is being assessed: "baseline" and "immediately after the completion" (2 months)
  Fried Frailty Phenotype (score)
Walking | Change is being assessed: "baseline" and "immediately after the completion" (2 months)
  Timed up and go test (seconds)
Strength | Change is being assessed: "baseline" and "immediately after the completion" (2 months)
  Grip strength by dynamometer (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Kwan, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- Pok Oi Hospital Neighbourhood Elderly Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruan Q, Yu Z, Chen M, Bao Z, Li J, He W. Cognitive frailty, a novel target for the prevention of elderly dependency. Ageing Res Rev. 2015 Mar;20:1-10. doi: 10.1016/j.arr.2014.12.004. Epub 2014 Dec 30. PMID 25555677
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Rosanna Chau MW, Chan SP, Wong YW, Lau MYP. Reliability and validity of the Modified Functional Ambulation Classification in patients with hip fracture. Hong Kong Physiotherapy Journal. 2013;31(1):41-44.
- [Background] Kelaiditi E, Cesari M, Canevelli M, van Kan GA, Ousset PJ, Gillette-Guyonnet S, Ritz P, Duveau F, Soto ME, Provencher V, Nourhashemi F, Salva A, Robert P, Andrieu S, Rolland Y, Touchon J, Fitten JL, Vellas B; IANA/IAGG. Cognitive frailty: rational and definition from an (I.A.N.A./I.A.G.G.) international consensus group. J Nutr Health Aging. 2013 Sep;17(9):726-34. doi: 10.1007/s12603-013-0367-2. PMID 24154642
- [Background] Desjardins-Crepeau L, Berryman N, Fraser SA, Vu TT, Kergoat MJ, Li KZ, Bosquet L, Bherer L. Effects of combined physical and cognitive training on fitness and neuropsychological outcomes in healthy older adults. Clin Interv Aging. 2016 Sep 19;11:1287-1299. doi: 10.2147/cia.s115711. eCollection 2016. PMID 27698558
- [Background] Lauenroth A, Ioannidis AE, Teichmann B. Influence of combined physical and cognitive training on cognition: a systematic review. BMC Geriatr. 2016 Jul 18;16:141. doi: 10.1186/s12877-016-0315-1. PMID 27431673
- [Background] Tait JL, Duckham RL, Milte CM, Main LC, Daly RM. Influence of Sequential vs. Simultaneous Dual-Task Exercise Training on Cognitive Function in Older Adults. Front Aging Neurosci. 2017 Nov 7;9:368. doi: 10.3389/fnagi.2017.00368. eCollection 2017. PMID 29163146
- [Background] de Vries AW, Faber G, Jonkers I, Van Dieen JH, Verschueren SMP. Virtual reality balance training for elderly: Similar skiing games elicit different challenges in balance training. Gait Posture. 2018 Jan;59:111-116. doi: 10.1016/j.gaitpost.2017.10.006. Epub 2017 Oct 5. PMID 29028622
- [Derived] Kwan RYC, Liu JYW, Fong KNK, Qin J, Leung PK, Sin OSK, Hon PY, Suen LW, Tse MK, Lai CK. Feasibility and Effects of Virtual Reality Motor-Cognitive Training in Community-Dwelling Older People With Cognitive Frailty: Pilot Randomized Controlled Trial. JMIR Serious Games. 2021 Aug 6;9(3):e28400. doi: 10.2196/28400. PMID 34383662